CLINICAL TRIAL: NCT01628770
Title: Iron Isomaltoside 1000 (Monofer)
Brief Title: Use of Iron Isomaltoside 1000 (Monofer) in Postpartum Anemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Nazli Hossain, Professor, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 7865
Record Dates: First submitted 2012-06-21; First posted 2012-06-27 (Estimated); Last update posted 2016-08-03 (Estimated); Status verified 2016-08

CONDITIONS: Postpartum Anemia
Keywords: iron; monofer; Pakistan
MeSH Terms: interventions — iron isomaltoside 1000; ferrous sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- parenteral iron (Experimental): dose will be calculated according to Ganzoni's formula, and will be administered by intravenous infusion
  Interventions: Drug: Iron isomaltoside 1000
- oral iron (Active Comparator): oral iron in form of ferrous sulphate 200 mg twice daily
  Interventions: Drug: Ferrous sulphate

INTERVENTIONS:
Drug: Iron isomaltoside 1000 — Iron molecule iron isomaltoside 1000 (Monofer) have been introduced in the market, which can be given in intravenous infusion forms, in a relatively short period of time, in a single setting, after calculation of the required dose. It can be given in a dose of 20mg/kg body weight.
  Other Names: Monofer
  Arms: parenteral iron
Drug: Ferrous sulphate — 200mg twice daily
  Arms: oral iron

SUMMARY:
The investigators hypothesized that both isomaltoside 1000 (Monofer), and oral iron preparation will be equally effective in correction of postpartum iron deficiency anemia.

DETAILED DESCRIPTION:
Iron molecule iron isomaltoside 1000 (Monofer) have been introduced in the market, which can be given in intravenous infusion forms, in a relatively short period of time, in a single setting, after calculation of the required dose. This preparation has been used for treatment of anemia in patients with chronic renal disease, gastrointestinal disorders, anemia of malignancy and in gynecological disorders. It does not require a test dose to be given before total dose, nor does it require any premedication. It can be given in a dose of 20mg/kg. The drug has been licensed for use in Europe in 2009. It has been used for treatment of anemia in patients with chronic renal disease, inflammatory bowel disease and in anemia due to malignancies

ELIGIBILITY:
Inclusion Criteria:

* Women within 24-48 hours of delivery with hemoglobin concentration < 10gm/dl

Exclusion Criteria:

* History of PPH, or significant blood loss in last 24 hours
* History of allergy to iron preparation
* Hemoglobin < 7gm/dl.
* Sign & symptoms of cardiac failure
* H/o blood transfusion in last 3 months
* H/O Chronic liver diseases.
* ↑ Creatinine > 2mg/dl.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 271 (Actual)
Dates: Start 2012-05; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
To see the rise in hemoglobin concentration of 2gm/dl or more. | 3 months
  To see the rise in hemoglobin concentration of 2gm/dl or more.This rise in hemoglobin concentration will be measured at day 14 and at 3 months, in both groups.

SECONDARY OUTCOMES:
secondary - time required for rise in hemoglobin concentration | 3 months
  time required for rise in hemoglobin concentration. Both groups will be compared in terms of time interval, to see the rise in hemoglobin concentration.

CONTACTS AND LOCATIONS:
Locations (1):
- Dow University of Health Sciences, Karachi, Sindh, Pakistan

REFERENCES:
- [Derived] Holm C, Thomsen LL, Langhoff-Roos J. Intravenous iron isomaltoside treatment of women suffering from severe fatigue after postpartum hemorrhage. J Matern Fetal Neonatal Med. 2019 Sep;32(17):2797-2804. doi: 10.1080/14767058.2018.1449205. Epub 2018 Mar 20. PMID 29558233